CLINICAL TRIAL: NCT04159246
Title: Role OF OCT-A TO Detect Possible Retinal Vascular Complications of Sofosbuvir (Sovaldi) in Patients With Hepatitis C Virus Infection
Brief Title: Role OF OCT-A TO Detect Possible Retinal Vascular Complications of Sofosbuvir in Patients With Hepatitis C
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Mohamed Saad (Other)
Responsible Party: Sponsor-Investigator, Mohamed Saad, Resident of Ophthalmology , Cairo University - researcher, Cairo University
Organization: Cairo University (Other)
Other Study IDs: s-5-2019
Record Dates: First submitted 2019-11-01; First posted 2019-11-12 (Actual); Last update posted 2019-11-12 (Actual); Status verified 2019-11

CONDITIONS: HCV Infection
MeSH Terms: conditions — Hepatitis C | interventions — Sofosbuvir

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Sovaldi group: patients with a documented diagnosis of chronic hepatitis C , normal renal functions And Rheumatoid factor tests (to exclude Purtscher like retinopathy as a rare presentation of cryoglobuinemia which considered one of extra hepatic manifestations of HCV)
  Interventions: Device: Optical coherence tomography angiography; Drug: Sofosbuvir (Sovaldi)

INTERVENTIONS:
Device: Optical coherence tomography angiography — Recent Optical coherence tomography angiography "OCT-A" will be performed to all patients before Treatment Administration.
  * Examination will be performed using Optovue AngioVue® "Optovue, Inc., Fremont, CA", which uses split-spectrum amplitude-decorrelation angiography algorithm, which minimizes motion noise. This system also allows quantitative analysis, since it provides numerical data about flow area and flow density maps.
  * The patient will be examined before and after finishing the treatment course
  Other Names: OCTA
Drug: Sofosbuvir (Sovaldi) — Sofosbuvir (tradename Sovaldi) is a direct acting antiviral medication used as part of combination therapy to treat chronic Hepatitis C , here it's used with Daclatasvir for 3 months
  Other Names: Sovaldi

SUMMARY:
The purpose of this study is to prospectively evaluate the value of Optical coherence tomography angiography (OCT-A) for the of detection of suspected retinal complications With Sofosbuvir (Sovaldi) in Patients With Hepatitis C Virus Infection

DETAILED DESCRIPTION:
During 3 months duration ( the treatment course duration) , Optical coherence tomography angiography (OCT-A) will be performed to 30 eyes of 30 patients with a documented diagnosis of chronic hepatitis C before and after receiving dual-therapy planning (Daclatasvir - Sofosbuvir (Sovaldi)) , normal renal functions And Rheumatoid factor tests , will undergo a comprehensive ophthalmic examination including:

* Manifest refraction
* Corrected distance visual acuity
* Anterior segment examination using slit lamp and tear film breakup time test
* Fundus examination

Recent Optical coherence tomography angiography (OCT-A) will be performed to all patients before Treatment Administration.

Examination will be performed using "Optovue AngioVue®" "Optovue, Inc., Fremont, CA", which uses split-spectrum amplitude-decorrelation angiography algorithm, which minimizes motion noise. This system also allows quantitative analysis, since it provides numerical data about flow area and flow density maps.

The patient will be examined before and after finishing the treatment course

* Optical coherence tomography angiography (OCT-A) image acquisition OCT-A will be done for all patients who are instructed to focus on a fixation target. OCTA images are obtained using the "RTVue XR Avanti (AngioVue; Optovue Inc, Fremont, California, USA)" machine and the incorporated "AngioVue OCT-A" system. Algorithm used is Split-Spectrum Amplitude Decorrelation Algorithm (SSADA). The scans which will be included in the study are of high signal strength more than 0.7 and they will be carefully inspected for motion artifacts. Automatic segmentation of intraretinal layers will be done using the automated software of the machine (version 2016.2.0; Optovue Inc). Angio-retina scan sizes in this study will be 6 X 6 mm for all eyes. Assessment of the macular vessel density will be done for superficial vascular layer, capillary plexus, deep capillary plexus and all retinal plexuses). Assessment of the foveal avascular zone on both superficial vascular layer (SVL) and deep capillary plexuses (DCP); including its size, perimeter and circularity (regularity) index. Circularity index is a measure of compactness of a shape relative to a circle. The circularity index of a circle is 1.0. Thus, a ratio closer to 0 indicates an irregular shape, and that closer to 1.0 indicates a circular shape.

All results will be in numerical values (percentage) to compare retinal vascularity before and after using the drug. Best corrected visual acuity (in values from o.o5 to 1.0) , dryness (in seconds) will be also measured before and after drug administration and it will be compared .

ELIGIBILITY:
Inclusion Criteria:

* Age between 20 and 80 years.
* Patients with chronic hepatitis C enrolled for (Daclatasvir - Sofosbuvir (Sovaldi)) .
* Patients who have normal ocular and fundoscopic examination before the onset of treatment.

Exclusion Criteria:

* Relapsed cases who have formerly taken the antiviral therapy (depending on the basis of medical record and filing system), or treated with interferon for any other cause .
* Patients with elevated renal functions or positive Rheumatoid factor (as a clue to diagnose Purtscher like retinopathy which is a rare presentation of cryoglobulinemia ,considered one of extra hepatic manifestations of HCV )

Ages: 20 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Convenience sample 30 eyes of 30 patients with a documented diagnosis of chronic hepatitis C
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2019-02-10 (Actual); Primary Completion 2019-11-30 (Estimated); Study Completion 2019-11-30 (Estimated)

PRIMARY OUTCOMES:
Assessment percentage of change in macular vessels density using OCTA | 3 months
  Evaluate the suspected retinal vascular complications With Sofosbuvir (Sovaldi) ) in Patients With Hepatitis C Virus Infection, All results will be in numerical values (percentage) to compare retinal vascularity before and after using the drug..
visual acuity changes with Sofosbuvir | 3 months
  Comparing best corrected visual acuity (in values from o.o5 to 1.0) before and after drug administration .

SECONDARY OUTCOMES:
amount of ocular dryness with Sofosbuvir using tear up breaking test | 3 months
  Measuring amount of ocular dryness using Tear-up breaking test, dryness will be evaluated in seconds before and after drug administration and it will be compared .
Role of Optical coherence tomography angiography (OCTA) in detection early signs retinopathy depending on changes in vascular density | 3 months
  Confirm the advantages of Optical coherence tomography angiography (OCT - A) in detection early signs retinopathy depending on changes in vascular density (evaluated as a percentage)
amount of ocular dryness with Sofosbuvir using Schirmer's | 3 months
  Measuring amount of ocular dryness using Tear-up breaking test, dryness will be evaluated in millimeters of wetness of schirmer's strips before and after drug administration and it will be compared .

CONTACTS AND LOCATIONS:
Overall Officials: Hany E Elmekewy, MD, Principal Investigator — Cairo University; Magada S Abdelaziz, MD, Principal Investigator — Cairo University; Yomna A Abdelwahab, MD, Principal Investigator — Cairo University; Mai I Mehrez, MD, Study Chair — National Hepatology & Tropical Medicine Research Institute
Locations (1):
- Cairo University - Kasr Alainy, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
All required non private data
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 30 November 2019
Access Criteria: upon request of Any qualified and specialized Doctor or medical journal

REFERENCES:
- [Background] Chebil A, Mammouri R, Abdallah MB, El Matri L. Purtscher-like Retinopathy as a Rare Presentation of Cryoglobulinemia. Middle East Afr J Ophthalmol. 2016 Apr-Jun;23(2):219-21. doi: 10.4103/0974-9233.177409. PMID 27162457
- [Background] Salman AG. Ocular Surface Changes With Sofosbuvir in Egyptian Patients With Hepatitis C Virus Infection. Cornea. 2016 Mar;35(3):323-8. doi: 10.1097/ICO.0000000000000736. PMID 26764884
- [Background] Manoharan N, Subramanian PS. A case of non-arteritic anterior ischemic optic neuropathy after completion of Harvoni therapy. Am J Ophthalmol Case Rep. 2017 Mar 8;6:55-57. doi: 10.1016/j.ajoc.2017.03.002. eCollection 2017 Jun. PMID 29260058
- [Background] Chin Loy K, Galaydh F, Shaikh S. Correction: Retinopathy and Uveitis Associated with Sofosbuvir Therapy for Chronic Hepatitis C Infection. Cureus. 2016 Jul 14;8(7):c3. doi: 10.7759/cureus.c3. PMID 27610281
- [Background] Lawitz E, Mangia A, Wyles D, Rodriguez-Torres M, Hassanein T, Gordon SC, Schultz M, Davis MN, Kayali Z, Reddy KR, Jacobson IM, Kowdley KV, Nyberg L, Subramanian GM, Hyland RH, Arterburn S, Jiang D, McNally J, Brainard D, Symonds WT, McHutchison JG, Sheikh AM, Younossi Z, Gane EJ. Sofosbuvir for previously untreated chronic hepatitis C infection. N Engl J Med. 2013 May 16;368(20):1878-87. doi: 10.1056/NEJMoa1214853. Epub 2013 Apr 23. PMID 23607594

DOCUMENTS (2):
  • Informed Consent Form (2019-08-15): https://cdn.clinicaltrials.gov/large-docs/46/NCT04159246/ICF_000.pdf
  • Study Protocol (2019-08-15): https://cdn.clinicaltrials.gov/large-docs/46/NCT04159246/Prot_001.pdf